CLINICAL TRIAL: NCT05367193
Title: Surgical Outcomes and Intraoperative Parameters Evaluation of 3D Visualization System for Vitreoretinal Diseases in Highly Myopic Eyes
Brief Title: 3D Visualization System for Vitreoretinal Diseases in Highly Myopic Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202110065DINC
Record Dates: First submitted 2022-04-26; First posted 2022-05-10 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2021-11

CONDITIONS: Patients With Highly Myopic Eyes
Keywords: vitreoretinal surgery; high myopia; Pars plana vitrectomy; 3D visualization system

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pars plana vitrectomy performed using NGENUITY® 3D Visualization System (Alcon, TX, USA) (Experimental): NGENUITY® 3D Visualization System (Alcon, TX, USA)
  Interventions: Procedure: pars plana vitrectomy; Device: NGENUITY® 3D Visualization System (Alcon, TX, USA)
- standard binocular microscope pars plana vitrectomy (Active Comparator): standard binocular microscope pars plana vitrectomy
  Interventions: Procedure: pars plana vitrectomy

INTERVENTIONS:
Procedure: pars plana vitrectomy — pars plana vitrectomy for vitreoretinal disease in highly myopic eyes
Device: NGENUITY® 3D Visualization System (Alcon, TX, USA) — Injection of ICG to stain internal limiting membrane
  Arms: pars plana vitrectomy performed using NGENUITY® 3D Visualization System (Alcon, TX, USA)

SUMMARY:
To investigate the surgical outcomes and intraoperative parameters evaluation of 3D visualization system for vitreoretinal diseases in highly myopic eyes

DETAILED DESCRIPTION:
The investigators aimed to compare the safety and efficacy of NGENUITY® 3D Visualization System (Alcon, TX, USA) in vitreoretinal surgery of highly myopic patients with standard binocular microscope pars plana vitrectomy of highly myopic patients. This is a randomized controlled study and will enroll highly myopic patients who had axial length more than 26 mm and needed vitreoretinal surgery. The enrolled patients will be randomized into "NGENUITY® 3D Visualization System (Alcon, TX, USA) group"(trial group) and "standard binocular microscope pars plana vitrectomy group"(controlled group). The investigators will compare the number of injections of dye (indocyanine green (ICG) or brilliant blue G (BBG)), total surgical time, total peeling time, exposure time of dye, power of endoilluminator, the rate of probe bending, surgical time, postoperative intraocular pressure (IOP), the rate of wound leakage, hypotony, subconjunctival hemorrhage, vitreous hemorrhage, retinal hemorrhage, and endophthalmitis, best-corrected visual acuity (BCVA), structural changes shown on OCT and so on between the two groups.

ELIGIBILITY:
Inclusion criteria:

1. Highly myopic patients (axial length ≥ 26mm, no upper limit)
2. Patient with vitreoretinal pathology that require vitrectomy who had not received previous ICG or BBG-assisted membrane peeling
3. Patient aged ≥ 20 years

Exclusion criteria:

1. Patient who had previous ICG or BBG-assisted membrane peeling
2. Patient who received combined vitrectomy and trabeculectomy
3. Patient with endophthalmitis or intraocular foreign body

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Number of injections of ICG | operation day
  Fixed and minimal concentration: ICG (25mg/vial) is diluted to 0.05% Fixed time: Each injection is 15 sec Interval time for washout: consistent as 10 sec

SECONDARY OUTCOMES:
Total surgical time | Intraoperative
  Total surgical time
ILM peeling time | operation day
  ILM peeling time
ICG exposure time | operation day
  ICG exposure time

CONTACTS AND LOCATIONS:
Overall Officials: Ho Tzyy-Chang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Data may be provided under reasonable request.